CLINICAL TRIAL: NCT00453726
Title: Evaluation of BNP in Patients With Severe Acute Respiratory Failure Requiring Non Invasive Mechanical Ventilation
Brief Title: Brain Natriuretic Peptide (BNP) Levels in Patients in Non Invasive Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Ospedale S. Giovanni Bosco (Other)
Responsible Party: Giovanni Ferrari, ASL TO4 Ospedale S. Giovanni Bosco
Other Study IDs: gbosco3
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Respiratory Insufficiency
Keywords: Natriuretic peptide brain; Continuous positive airway pressure; Intermittent positive pressure breathing; Respiratory insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Non invasive mechanical ventilation

SUMMARY:
The purpose of the study is to evaluate variation of BNP in non invasive mechanical ventilated patients with severe acute respiratory failure.

DETAILED DESCRIPTION:
The aim of the study is to evaluate in patients with severe acute respiratory failure requiring non invasive mechanical ventilation BNP levels at admission and during the following 24 hours during non invasive mechanical ventilation (Non Invasive Positive Pressure Ventilation or Continuous positive airway pressure).

Because in patients affected by acute respiratory failure it is often difficult to distinguish if the disease precipitating the respiratory failure is a cardiac disease or a lung disease, aim of the present study is to evaluate the discriminating role that BNP could have in this group of patients; evaluation will be completed, once obtained clinical stabilisation, with an echocardiography and respiratory functional test.

ELIGIBILITY:
Inclusion Criteria:

* Severe respiratory distress (use of respiratory accessory muscles);
* Respiratory rate > 25 per minute;
* Respiratory acidosis (pH < 7.35 and PaCO2 > 45 mmHg);
* PaO2/FiO2 < 250

Exclusion Criteria:

* Age < 18 years;
* Facial deformities;
* Pneumothorax;
* Shock or systolic arterial pressure below 90 mmHg with amine infusion;
* Life-threatening arrhythmias;
* Need for immediate endotracheal intubation (PaO2/FiO2 < 100 with FiO2 100%, respiratory rate < 10, GCS < 8);
* Lack of co-operation from the patient;
* Recent esophageal-gastric surgery;
* Inability to clear secretions;
* Drugs that may interfere with BNP secretion;
* Severe obesity;
* Hepatic cirrhosis with ascitis;
* Endocrine disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the city of Torino, admitted to the emergency department for acute respiratory failure.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-05; Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ferrari, MD, Principal Investigator — Ospedale San Giovanni Bosco ASL4 Torino Italy
Locations (1):
- Ospedale San Giovanni Bosco Medicina d'Urgenza, Turin, Piedmont, Italy